CLINICAL TRIAL: NCT05832840
Title: Validation of a Survey Instrument for Screening of Pre-Pregnant Women - The PREPSA SCALE
Brief Title: Survey Tool for Screening of Anemia in Women Before Pregnancy
Acronym: PREPSA
Status: Completed | Type: Observational
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Thomas Jefferson University (Other); Jawaharlal Nehru Medical College (Other); RTI International (Other)
Responsible Party: Sponsor
Other Study IDs: GN08 PREPSA
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Anemia Complicating Pregnancy; Anemia Complicating Childbirth; Anemia Complicating the Puerperium
Keywords: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational and cross-sectional study is to develop and validate a survey that can be used to identify anemia, and its severity, among pre-pregnant women allowing for the timely implementation of focused public health and personalized interventions.

Participants will be asked 26 survey questions about menstrual history and provide a 5 ml venous blood sample to measure hemoglobin, ferritin, and transferrin saturation levels.

DETAILED DESCRIPTION:
Despite a variety of governmental campaigns and funded programs, anemia rates among reproductive age women in low- and middle-income countries (LMICs) have not decreased over the past few decades. Iron deficiency is associated with increases in morbidity and mortality in both non-pregnant and pregnant women, as well as their offspring.

Up to 500 currently married women between 18 and 25 years old who are not pregnant, have never been pregnant, and are not using any type of contraception other than barrier methods will be recruited for this study from primary health centres (PHCs) in Belagavi , Karnataka, India.

Accredited Social Health Activists (ASHAs) will identify potentially eligible participants and bring them to participating primary healthcare centers (PHCs) for screening, consent, and enrollment. Once enrolled, trained female interviewers will administer the PREPSA survey to the participant and a laboratory technician will draw a blood sample (upon completion of the survey or within four weeks) to analyze hemoglobin, ferritin, and transferrin saturation values. The survey responses that most closely align with low iron indices will be identified and become the basis of a scored, validated instrument which may be weighted based upon the strength of the associations found. Results will inform future health outcome trials.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 25 year old women
* Not currently pregnant and have never been pregnant
* Currently married
* If last menstrual period >6 weeks ago, exclude pregnancy via pregnancy test

Exclusion Criteria:

* Currently using any form of contraception other than barrier methods

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Currently married pre-pregnant women (n=500), ages 18-25 years, in Belagavi, Karnataka, India
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Validation of survey instrument | Up to four weeks following pre-pregnancy administration of PREPSA scale
  The PREPSA Scale will be administered to pre-pregnant women and a blood draw within four weeks will be used to assess anemia status and support validation of the PREPSA Scale. The minimum value on the scale is a score of zero. The maximum value on the scale is a score of forty. This is based on the number of items plus the value of the highest coded category on items with more than one category. A higher score means a worse outcome and is associated with higher levels of iron deficient anemia.

CONTACTS AND LOCATIONS:
Locations (1):
- Jawaharlal Nehru Medical College, Belagavi, India

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available through the NICHD Data and Specimen Hub (N-DASH system, a publicly accessible online archive, following publication of the primary paper.
Supporting Information: Study Protocol, SAP
Time Frame: No more than one year after publication of the primary paper. No end date.
Access Criteria: Access will follow procedures in accordance with those outlined by the NICHD Data and Specimen Hub (N-DASH).